CLINICAL TRIAL: NCT04551040
Title: Assessing Target Engagement of Terazosin in Healthy Adults
Brief Title: Target Engagement of Terazosin in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Jordan Schultz, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202005461
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Terazosin; Hytrin; Target engagement; Glycolysis; ATP
MeSH Terms: interventions — Terazosin

STUDY DESIGN:
Intervention Model Description: Single group of healthy older adults
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary Cohort (Experimental): Titrating doses of terazosin starting at 1mg daily and increasing to 5mg daily on a weekly basis for five weeks.
  Interventions: Drug: Terazosin

INTERVENTIONS:
Drug: Terazosin — Terazosin 1 mg oral capsule
  Other Names: Hytrin

SUMMARY:
The purpose of the study is to assess the target engagement of Terazosin (TZ) in a single cohort of 6 healthy adult participants. During the study participants will undergo PET/CT scans, 7-Tesla MRI scans, blood draws, and an optional lumbar puncture (LP.)

DETAILED DESCRIPTION:
The study is a single center, 37-day, controlled pilot study to assess the target engagement of Terazosin (TZ) in a single cohort of 6 healthy adult participants (3 men and 3 women.) During the study participants will undergo PET/CT scans, 7-Tesla MRI scans, blood draws, and an optional lumbar puncture (LP.) Participants will have their baseline ATP levels measured (at 0mg TZ.) They will then take doses of TZ at 1mg and will increase their dose on a weekly basis by 1mg until they reach a total dose of 5mg. ATP levels will be assessed on study days 8 and 36. Participants interested in voluntarily donating a sample of cerebral spinal fluid will undergo an optional lumbar puncture on study day 37.

The purpose of the study is to gain a better understanding of the mechanisms in which TZ acts in the brain. TZ was recently discovered to increase energy levels (in the form of ATP molecules) in the brain by enhancing glycolysis. By using different brain imaging techniques, blood assays and cerebral spinal fluid assays, the study will attempt to: 1) quantify the rate of glycolysis in the brain at different dosages of TZ, 2) quantify ATP levels in the brain at different dosages of TZ, 3) quantify ATP levels in blood at different dosages of TZ, and 4) assess the brain permeability of TZ. It is hoped that knowledge gained from the study will help guide future clinical trials using TZ for the treatment of various neurodegenerative diseases such as Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men or women aged 60-90

Exclusion Criteria:

* History of stroke
* Ineligibility for MRI (e.g. soft tissue metallic implants, clips, cardiac pacemaker, cardiac defibrillator, internal pacing wires, metallic fragments, shrapnel, etc.)
* Current use of more than one of the following classes of medications: beta blockers, ace inhibitors, angiotensin receptor blockers, calcium channel blockers, or diuretics
* Use of any alpha blockers (terazosin, doxazosin, alfuzosin, prazosin, or tamsulosin) in the past year.
* Current use of the over-the-counter supplement yohimbe
* Orthostatic hypotension defined as symptomatic decrease in BP > 20mmHg systolic or > 10mmHg diastolic and HR increase < 20bpm on supine to sitting or standing.
* Alcohol and drug abuse
* Clinically significant traumatic brain injury
* History of Type I diabetes
* Uncontrolled Type II diabetes
* Other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study or increase fall risk
* Use of investigational drugs within 30 days before screening
* History of hemodynamic instability
* For females: pregnancy or breastfeeding

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of glycolysis in the brain at baseline | Study day 1
  Use of FDG PET to quantify glycolysis in the brain at baseline prior to initiation of terazosin
Change in glycolysis in the brain from baseline to 1 week (1mg of terazosin) | Study day 8
  Use of FDG PET to determine how TZ quantitatively increases glycolysis as measured by FDG uptake from baseline to 1 week (Day 8/ 1mg TZ)
Change in glycolysis in the brain from baseline to 5 weeks (5mg of terazosin) | Study day 36
  Use of FDG PET to determine how TZ quantitatively increases glycolysis as measured by FDG uptake from baseline to 5 weeks (Day 36/ 5mg TZ)
Quantification of ATP in brain at baseline | Study day 1
  Use of Magnetic Resonance Spectroscopy (MRS) to quantify ATP in the brain at baseline prior to initiation of terazosin
Change in ATP in the brain from baseline to 1 week (1mg of terazosin) | Study day 8
  Use of Magnetic Resonance Spectroscopy (MRS) determine how TZ quantitatively increases ATP as measured by MRS from baseline to 1 week (Day 8/ 1mg TZ)
Change in ATP in the brain from baseline to 5 weeks (5mg of terazosin) | Study day 36
  Use of Magnetic Resonance Spectroscopy (MRS) determine how TZ quantitatively increases ATP as measured by MRS from baseline to 5 weeks (Day 36/ 5mg TZ)
Quantification of ATP in blood at baseline | Study day 1
  Use of a novel assay to quantify ATP in the blood at baseline prior to initiation of terazosin
Change in ATP in the blood from baseline to 1 week (1mg of terazosin) | Study day 8
  Use of a novel assay to determine how TZ quantitatively increases ATP in the blood from baseline to 1 week (Day 8/ 1mg TZ)
Change in ATP in the blood from baseline to 5 week (1mg of terazosin) | Study day 36
  Use of a novel assay to determine how TZ quantitatively increases ATP in the blood from baseline to 5 weeks (Day 36/ 5mg TZ)
Quantification of TZ in Cerebrospinal Fluid | Study day 37
  Participants will be given the option to undergo a lumbar puncture on Day 37 (5 mg TZ). Their blood will also be drawn to compare levels of TZ in the blood to levels detected in the CSF.

SECONDARY OUTCOMES:
Safety and Tolerability | Ongoing (days 1 - 37)
  We will assess patient-reported adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Schultz, PharmD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
The Michael J. Fox Foundation for Parkinson's Research requires all funded investigators to share data with the foundation. The Foundation will make de-identified, patient-specific data available to interested investigators upon reasonable request.

REFERENCES:
- [Background] Chen X, Zhao C, Li X, Wang T, Li Y, Cao C, Ding Y, Dong M, Finci L, Wang JH, Li X, Liu L. Terazosin activates Pgk1 and Hsp90 to promote stress resistance. Nat Chem Biol. 2015 Jan;11(1):19-25. doi: 10.1038/nchembio.1657. Epub 2014 Nov 10. PMID 25383758
- [Background] Cai R, Zhang Y, Simmering JE, Schultz JL, Li Y, Fernandez-Carasa I, Consiglio A, Raya A, Polgreen PM, Narayanan NS, Yuan Y, Chen Z, Su W, Han Y, Zhao C, Gao L, Ji X, Welsh MJ, Liu L. Enhancing glycolysis attenuates Parkinson's disease progression in models and clinical databases. J Clin Invest. 2019 Oct 1;129(10):4539-4549. doi: 10.1172/JCI129987. PMID 31524631
- [Background] Schapira AH. Mitochondria in the aetiology and pathogenesis of Parkinson's disease. Lancet Neurol. 2008 Jan;7(1):97-109. doi: 10.1016/S1474-4422(07)70327-7. PMID 18093566
- [Background] Hoyer S. Brain glucose and energy metabolism during normal aging. Aging (Milano). 1990 Sep;2(3):245-58. doi: 10.1007/BF03323925. PMID 1982730
- [Background] Cunnane S, Nugent S, Roy M, Courchesne-Loyer A, Croteau E, Tremblay S, Castellano A, Pifferi F, Bocti C, Paquet N, Begdouri H, Bentourkia M, Turcotte E, Allard M, Barberger-Gateau P, Fulop T, Rapoport SI. Brain fuel metabolism, aging, and Alzheimer's disease. Nutrition. 2011 Jan;27(1):3-20. doi: 10.1016/j.nut.2010.07.021. Epub 2010 Oct 29. PMID 21035308
- [Background] Blesa J, Phani S, Jackson-Lewis V, Przedborski S. Classic and new animal models of Parkinson's disease. J Biomed Biotechnol. 2012;2012:845618. doi: 10.1155/2012/845618. Epub 2012 Mar 28. PMID 22536024
- [Background] Hoffe B, Holahan MR. The Use of Pigs as a Translational Model for Studying Neurodegenerative Diseases. Front Physiol. 2019 Jul 10;10:838. doi: 10.3389/fphys.2019.00838. eCollection 2019. PMID 31354509
- [Background] Hoegger MJ, Fischer AJ, McMenimen JD, Ostedgaard LS, Tucker AJ, Awadalla MA, Moninger TO, Michalski AS, Hoffman EA, Zabner J, Stoltz DA, Welsh MJ. Impaired mucus detachment disrupts mucociliary transport in a piglet model of cystic fibrosis. Science. 2014 Aug 15;345(6198):818-22. doi: 10.1126/science.1255825. PMID 25124441
- [Background] Rogers CS, Stoltz DA, Meyerholz DK, Ostedgaard LS, Rokhlina T, Taft PJ, Rogan MP, Pezzulo AA, Karp PH, Itani OA, Kabel AC, Wohlford-Lenane CL, Davis GJ, Hanfland RA, Smith TL, Samuel M, Wax D, Murphy CN, Rieke A, Whitworth K, Uc A, Starner TD, Brogden KA, Shilyansky J, McCray PB Jr, Zabner J, Prather RS, Welsh MJ. Disruption of the CFTR gene produces a model of cystic fibrosis in newborn pigs. Science. 2008 Sep 26;321(5897):1837-41. doi: 10.1126/science.1163600. PMID 18818360
- [Background] Hytrin (terazosin) [package insert]. Abbott Indistries, North Chicago, IL. 2001.
- [Background] Matthews DC, Lerman H, Lukic A, Andrews RD, Mirelman A, Wernick MN, Giladi N, Strother SC, Evans KC, Cedarbaum JM, Even-Sapir E. FDG PET Parkinson's disease-related pattern as a biomarker for clinical trials in early stage disease. Neuroimage Clin. 2018 Aug 10;20:572-579. doi: 10.1016/j.nicl.2018.08.006. eCollection 2018. PMID 30186761
- [Background] Patel A, Malinovska L, Saha S, Wang J, Alberti S, Krishnan Y, Hyman AA. ATP as a biological hydrotrope. Science. 2017 May 19;356(6339):753-756. doi: 10.1126/science.aaf6846. PMID 28522535
- [Background] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123